CLINICAL TRIAL: NCT03495843
Title: Assessing Normative Data, Reliability and the Influence of Body Position and Axial Load on Spinal Stiffness by Electromechanical Measurements in Young Healthy Adults
Brief Title: The Influence Body Position and Axial Load on Spinal Stiffness
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Swanenburg, PhD, Balgrist University Hospital
Other Study IDs: 2017-01245
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spinal stiffness — Spinal stiffness will be assessed with a device, which measures tissue compliance according to the concept of impulse-response

SUMMARY:
The objective of this study is to examine the influence of body position and additional axial load on spinal stiffness in young healthy adults.

DETAILED DESCRIPTION:
Spinal stiffness plays an important role in the assessment of the spine in the clinical daily routine. It is often performed as a manual PA-pressure test in the prone position. The spinal stiffness is the result of the resistance from the active, passive and neurological subsystems, like muscles (active), ligaments, joint capsule and the skin (passive). Further research had shown, that the spinal stiffness depends also from other factors. It is increased by axial compression. A better understanding of spinal stiffness leads to novel insights into spinal stabilization mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* Acute backpain (thoracal or lumbar)
* History of significant backpain (thoracal or lumbar) or radiating pain down the leg
* Contraindications to PA mobilisation/manipulation
* Spinal fractures
* Spinal tumors
* Surgical intervention in the thoracic and lumbar spine
* Local infections of the spine or the surrounding tissue

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Young healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Spinal stiffness | Day one of the study
  posterior-to-anterior spinal will be assesd in prone and upright body position and in upright body position with additional axial.
  The device measures tissue compliance according to the concept of impulse-response. A force of exact 80 Newton will be applied from the device to the process spinous. The expected impulse-response (result) will be between 40 Newton and 70 Newton.

SECONDARY OUTCOMES:
Pain during measuring spinal stiffness | Day one of the study
  Visual Analogue Pain Rating Scale will be used if the particepants feel any pain during the measurement.The participant will be asked to rate his pain intensity on a straight line (100 millimeter) with two endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No